CLINICAL TRIAL: NCT00555074
Title: Efficacy of Oral Sodium Tungstate (200 mg/Day)on Weight Loss in Subjects With Grade I-II Obesity
Brief Title: Sodium Tungstate in Obesity
Acronym: TROTA-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacio Clinic Barcelona (Other)
Responsible Party: Josep Vidal, Hospital Clinic Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TROTA-1; EudraCT: 2006-000567-28
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — sodium tungstate(VI)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sodium Tungstate
  Interventions: Drug: Sodium Tungstate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Tungstate — Sodium Tungstate, 200 mg BID, oral route during 6 weeks
  Arms: 1
Drug: Placebo — Placebo, BID, oral route during 6 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of sodium tungstate versus placebo in patients with obesity (grade I and II).

ELIGIBILITY:
Inclusion Criteria:

* BMI: 30-39.9 Kg/m2
* In case of male gender, 18 to 65 years old
* In case of female gender, diagnosis of menopause
* Body weight changes < 3 kg in the last 3 months
* In case of arterial hypertension or dyslipemia, no changes in dose in the last 2 months

Exclusion criteria:

* In case of female gender, absence of menopause
* Evidence of secondary causes of obesity
* Diabetes, type II
* Concomitant treatment with drugs affecting body weight
* Previous surgical intervention of obesity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
weight loss | six weeks

SECONDARY OUTCOMES:
changes in lipids | 6 weeks
changes in caloric intake and in hungry sensation | 6 weeks
resting metabolic rate | 6 weeks
changes in body composition | 6 weeks
adverse events | 6 weeks
changes in hormonal parameters | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Josep Vidal, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospiral Clinic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Hanzu F, Gomis R, Coves MJ, Viaplana J, Palomo M, Andreu A, Szpunar J, Vidal J. Proof-of-concept trial on the efficacy of sodium tungstate in human obesity. Diabetes Obes Metab. 2010 Nov;12(11):1013-8. doi: 10.1111/j.1463-1326.2010.01293.x. PMID 20880348